CLINICAL TRIAL: NCT05127668
Title: Assessment by Ultrasound of the Degree of Venous Dilation, Comparison Between Venodilation by Airglove (TM) Versus Warm-water Immersion (WWI)
Brief Title: Efficacy of AirGLovE in Difficult Venous Access
Acronym: EAGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HLS/PSWAHS/18/168
Record Dates: First submitted 2021-09-14; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cancer
Keywords: Cannulation,; Chemotherapy; Difficult venous access; Difficult venepuncture; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective cross-sectional comparative study
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and reviewer were masked to the results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airglove arm (Experimental): Participants on the airglove arm were subjected to warming of their forearms using the Airglove device at 38.5oC.
  Interventions: Device: Airglove (TM)
- Warm-water Immersion arm (Experimental): Participants on the WWI arm were subjected to warming by immersing their forearms into a bucket of warm water at 38.5oC.
  Interventions: Device: Warm-water Immersion

INTERVENTIONS:
Device: Airglove (TM) — A sterile polythene-balloon was inflated around the forearm using the AirGloveTM to 38.5oC at setting number-3 for 3 minutes, then removed and the degree of venodilation assessed by ultrasound.
  Arms: Airglove arm
Device: Warm-water Immersion — The upper limbs (to the level of mid-humerus) of participants were immersed in a container filled with a mix of cold-and warm tap-water to 38.5oC for 3 minutes in the WWI method. Arms were towel-dried, and the degree of venodilation was assessed by ultrasound
  Arms: Warm-water Immersion arm

SUMMARY:
To determine whether Airglove™ warming device dilates upper limb veins to the same degree as the warm water immersion (WWI) method.

DETAILED DESCRIPTION:
Failure to cannulate to gain intra-venous access is a common occurrence in patients undergoing chemotherapy, obese patients, intravenous drug users and those with chronic medical problems leading to peripheral venous collapse. Difficulty in gaining IV-access is a serious medical consequence since important life-saving drugs, fluids, blood transfusions, and other medication are usually given via the intravenous route. Most chemotherapy units in the UK rely on venous dilation by immersing the forearm of patients with "difficult to cannulate veins" (DTCV) into a bucket of warm water. There are however, limitations in this method such as controlling water temperature and ensuring proper sterility.

A new device Airglove™ has been developed which directs warm air over the forearm in a polythene sleeve causing venodilation. Preliminary studies in chemotherapy patients suggest that the Airglove™ causes venodilation to the extent of the warm water immersion technique, however further evidence is required with testing on normal healthy volunteers.

Aims and Objectives:

To determine whether Airglove™ warming device dilates upper limb veins to the same degree as the warm water immersion (WWI) method.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 18 years old
* Able to give written informed consent
* Able to understand and complete questionnaire forms independently

Exclusion Criteria:

* Participants < 18 years old
* Participants with cancer and/or undergoing chemotherapy
* Participants with difficult to cannulate veins (DTCV)
* Participants with lymphoedema in either hand
* Participants with pre-existing Raynaud's disease
* Participants with Diabetes (Type 1 & 2)
* Participants with generalised anxiety disorder
* Participants with diagnosis of hypertension
* Participants with any cardiovascular disease, previous stroke, episodes of DVT, recent treatment for venous thromboembolism (VTE), recently administered heparin, participants on warfarin or any anticoagulant treatment (including NOACs).
* Participants not able to give written informed consent
* Participants not able to comprehend or complete questionnaire forms independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Name of Measurement: Change in measurement of vein diameter by ultrasound | Change from baseline measurements taken within 2 minutes of the intervention
  MEASUREMENT TOOL: GE Logic S8 multi-frequency linear-array transducer (L6-15MHz), two-dimension B-mode ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Glasgow Calenonian University, Glasgow, South Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT05127668/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT05127668/SAP_001.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT05127668/ICF_002.pdf